CLINICAL TRIAL: NCT00375297
Title: Randomized Double Blind Placebo Controlled Study of Sildenafil for Treatment of Serotonergic Reuptake Inhibitor Associated Sexual Dysfunction in Women With Major Depression Treated to Remission
Brief Title: Study of Sildenafil for Treatment of SSRI-Antidepressant Sexual Dysfunction in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99321; Acc# 4-37011
Record Dates: First submitted 2005-09-11; First posted 2006-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Sexual Dysfunction; Depression
Keywords: antidepressants; sexual dysfunction; women; sildenafil; PDE5 inhibitors; serotonin reuptake inhibitor antidepressants
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Depression | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
This prospective double-blind, placebo-controlled (DBPC) study, assessed the efficacy of sildenafil in women with serotonin reuptake inhibitor antidepressant-associated sexual dysfunction (SRI-AASD) following the same protocol which previously established efficacy in men with SRI-AASD.

DETAILED DESCRIPTION:
This prospective double-blind, placebo-controlled (DBPC) study, assessed the efficacy of sildenafil in women with serotonin reuptake inhibitor antidepressant-associated sexual dysfunction (SRI-AASD) following the same protocol which previously established efficacy in men with SRI-AASD. Women (n=100) with MDD-remission and SRI-AASD were randomized to receive sildenafil (50-100mg) or placebo for 8 weeks, followed by 8-weeks open-label extension. Sexual function was assessed using the Clinical Global Impression-Sexual Function (CGI-SF), with positive response defined as a score <3, and UNM-SFI, ASEX, SFQ-FSD sexual function questionnaires. Depression was monitored using the HAM-D17. Hypothalamic-pituitary-adrenal-gonadal hormones were measured at baseline and DB-endpoint.

ELIGIBILITY:
Inclusion Criteria:S Subjects will be females only, ages 18 to 50 years.

* Subjects have been taking an SSRI, venlafaxine, nefazodone, or tri/hetero cyclic antidepressant for treatment of depression for at least 8 weeks, are currently at a stable dose of the antidepressant for at least 4 weeks, and have been consistently experiencing arousal dysfunction [inability to attain or maintain until completion of sexual activity an adequate lubrication swelling response of sexual excitement] or orgasmic dysfunction [delayed orgasm/anorgasmia following a normal sexual excitement phase] that interferes with sexual functioning for at least 4 weeks.
* Subjects must currently be euthymic (HAM-D<10) and without significant anxiety symptoms (HAM-A<10).
* Subjects must have had no sexual dysfunction prior to taking an antidepressant and there must be a clear temporal relationship of the sexual dysfunction to the antidepressant treatment. [Note - sexual dysfunction occurring as a symptom of the depressive disorder for which AD treatment was initiated is not considered to be a pre-existing condition in this definition].
* Subjects must meet at least one of the following criteria:

  1. Inability to have an orgasm (anorgasmia), according to patient opinion.
  2. Clinically significant orgasm delay with masturbation or intercourse that according to patient opinion:

     1. represents a meaningful delay compared with the subject's usual time to achieve orgasm in response to sexual stimulation prior to antidepressant medication and
     2. interferes with subject's sexual function.
  3. Inability to attain or maintain until completion of sexual activity an adequate lubrication swelling response of sexual excitement that according to patient opinion interferes with subject's sexual function compared to prior to antidepressant medication.
* Subjects must experience at least one of the above criterion items (#1-3) with distress and or disability.
* Subjects must be having or had been having some form of regular sexual activity (i.e., masturbation, oral sex, intercourse) at least twice monthly prior to the antidepressant treatment and are willing to continue efforts at sexual activity at least once weekly for the duration of the study.
* Subjects must be in good general physical health.
* Subjects must have given informed consent to participate in the study.

Exclusion Criteria:

* Primary or prior diagnosis of a sexual disorder (other than the side effect of the antidepressant drug or symptom of major depression).
* Vaginal, clitoral, or other sexual organ anatomical deformities.
* Post-hysterectomy with or without oophorectomy without at least six months of postoperative normal sexual function preceding depression and antidepressant treatment.
* Any uncontrolled psychiatric disorder.
* Alcohol or substance abuse or dependence within past twelve months.
* Using or likely to use any nitrate or nitric oxide donors in any form (oral, sublingual, buccal, transdermal, inhalational, or aerosol).
* Hamilton Depression and/or Anxiety Scale score [either] > 10.
* Blood pressure outside 90/50 or 170/100.
* Use of investigational drugs within prior 3 months or during study.
* Current use of other drugs for antidepressant induced sexual dysfunction.
* Hormone replacement therapy unless patient has been on stable dose of hormone therapy for at least 3 months prior to the antidepressant treatment and had no sexual dysfunction while on the same hormone therapy regimen, and there is no change in the hormone replacement therapy during the study.
* Pregnancy, lactating, or planning to become pregnant during the study.
* Child bearing potential subjects unwilling and/or not prepared and/or who are judged unreliable to use an acceptable and verifiable form of contraception during the study (these include IUD, double barrier or hormonal methods of birth control).
* Any clinically significant abnormality of the screening physical examination or safety laboratory test results.
* Subjects whose sexual partners are suffering from and/or receiving treatment for sexual dysfunction.
* eceiving psychosexual or other therapy for sexual dysfunction and not willing to discontinue that treatment at screening.
* Amenorrhea for greater than 1 year.
* Subjects whose sexual dysfunction is considered to be situational, i.e. limited to certain types of situations, stimulation, or partners.
* Subjects not attempting some form of regular sexual activity at least twice monthly and at least once weekly during study visit intervals for the duration of the entire study.
* Changes in antidepressant agent and or dose of prescribed antidepressant agent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2001-01; Study Completion 2005-06

PRIMARY OUTCOMES:
Clinical global improvement in sexual function

SECONDARY OUTCOMES:
UNM-Sexual function inventory
Arizona Sexual Function Scale
Female sexual function questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: George Nurnberg, MD, Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Nurnberg HG, Hensley PL, Gelenberg AJ, Fava M, Lauriello J, Paine S. Treatment of antidepressant-associated sexual dysfunction with sildenafil: a randomized controlled trial. JAMA. 2003 Jan 1;289(1):56-64. doi: 10.1001/jama.289.1.56. PMID 12503977
- [Derived] Nurnberg HG, Hensley PL, Heiman JR, Croft HA, Debattista C, Paine S. Sildenafil treatment of women with antidepressant-associated sexual dysfunction: a randomized controlled trial. JAMA. 2008 Jul 23;300(4):395-404. doi: 10.1001/jama.300.4.395. PMID 18647982